CLINICAL TRIAL: NCT06770764
Title: A Phase 1/1b, Multicenter, Open-label, Dose Escalation and Expansion Study Evaluating the Safety, Pharmacodynamics, and Pharmacokinetics of ODC-IL2 Administered Via Intravenous Infusion in Adult Patients With Advanced or Metastatic Solid Tumors
Brief Title: Dose Escalation and Expansion Study Evaluating ODC-IL2 in Adult Patients With Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Trutino Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TRT-ODC-IL2-001
Record Dates: First submitted 2025-01-02; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Advanced Solid Tumors; Metastatic Solid Tumors
Keywords: ODC-IL2; Tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ODC-IL2 monotherapy dose escalation (Experimental): All patients will receive ODC-IL2 as a single agent infused IV over 60 minutes on Days 1 and 15 of a 28 day cycle.
  Interventions: Drug: ODC-IL2
- ODC-IL2 monotherapy dose expansion (Experimental): All patients will receive ODC-IL2 as a single agent infused IV over 60 minutes on Days 1 and 15 of a 28 day cycle.
  Interventions: Drug: ODC-IL2

INTERVENTIONS:
Drug: ODC-IL2 — ODC-IL2 as a single agent infused IV over 60 minutes on Days 1 and 15 of a 28 day cycle.
  Other Names: Investigation product

SUMMARY:
This is a first-in-human, Phase I, multicenter, open-label, dose escalation study with dose expansion to evaluate the safety and antitumor activity of ODC-IL2 in patients with advanced or metastatic solid tumors. ODC-IL2 is a conditionally activated IL-2 prodrug and will be administered as a single agent via intravenous infusion on Days 1 and 15 of a 28-day cycle. Up to approximately 50 patients will be enrolled in this study.

DETAILED DESCRIPTION:
This is a first-in-human, Phase I, multicenter, open-label, dose-escalation and expansion study evaluating the safety, pharmacodynamics, pharmacokinetics and preliminary antitumor activity of ODC-IL2 for the treatment of patients with advanced or metastatic solid tumors. Part 1 of the study is dose escalation of ODC-IL2 and up to 18 to 30 patients (for up to 10 dose levels) or more will be enrolled in this portion of the study (depending on the number of dose escalation cohorts and patients per cohort required). Once the MTD or RDR has been established in dose escalation, a Part 2 expansion will begin. The dose-expansion cohort at a single dose level will enroll approximately 20 patients with advanced solid tumors to further evaluate safety and assess for signals of antitumor activity. The objective of the dose-escalation and expansion is to define, with a limited number of patients, the safety and toxicity characteristics of ODC-IL2. The study drug ODC-IL2 is a conditionally activated IL-2 prodrug and will be administered as a single agent by IV infusion over a 60-minute period on Days 1 and 15 of the treatment cycle. A treatment cycle is defined as 28 days.

This trial will enroll adult patients with advanced or metastatic solid tumors that have not responded to or have recurred following treatment with available therapies. Up to approximately 50 evaluable patients may be enrolled in this study across the dose-escalation and dose-expansion cohorts. Enrollment in this study is anticipated to be 15 to 18 months.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all the following criteria to participate in the study:

1. Histologically or cytologically confirmed advanced or metastatic solid tumors, for which no other standard treatment is available or appropriate, or for which the Trutino Biosciences Protocol #: TRT-ODC-IL2-001 Version: 1.0 Date: 20 September 2024 standard of care is refused by the patient due to tolerability or the Investigator believes the patient will not tolerate standard-of-care therapy
2. Advanced or metastatic tumors measurable per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria;
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
4. Life expectancy of at least 3 months;
5. Age ≥ 18 years;
6. Signed, written Institutional Review Board (IRB)/Ethics Committee (EC)-approved informed consent
7. Acceptable liver function:

   * Bilirubin ≤ 1.5 times upper limit of normal (ULN) or ≤ 5 × institutional ULN for patients who have serum bilirubin increases due to underlying Gilbert's Syndrome (familial benign unconjugated hyperbilirubinemia).
   * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase ≤ 2.5 x ULN (if liver metastases are present, then ≤ 5 x ULN is allowed)
8. Acceptable renal function:

   • Calculated creatinine clearance ≥ 50 mL/min using the Cockcroft-Gault equation.
9. Acceptable hematologic status:

   * Absolute neutrophil count ≥ 1500 cells/mm3
   * Platelet count ≥ 75,000 (plt/mm3)
   * Hemoglobin ≥ 9 g/dL
10. A negative serum pregnancy test (if a woman of childbearing potential);
11. Women of childbearing potential (WOCBP) and men with WOCBP partners must agree to use adequate contraception (hormonal method of birth control; intrauterine devices or abstinence) prior to study entry, for the duration of study participation and for 4 months after the last dose of study drug. Should a female trial participant or a female partner of a male trial participant become pregnant or suspect she is pregnant during the study, the Investigator must be informed immediately.

Exclusion Criteria:

1. New York Heart Association Class III or IV, cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, or evidence of ischemia on electrocardiogram (ECG)
2. Have a corrected QT interval (using Fridericia's correction formula) (QTcF) of > 470 msec
3. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
4. Known active brain metastases; patients with previously treated, clinically stable, radiologically stable brain metastases (without evidence of progression in 4 weeks) and without the requirement for treatment with corticosteroids in prior 3 weeks may be considered for enrollment after discussion with the Medical Monitor
5. History of prior organ transplant
6. Conditions requiring systemic treatment with corticosteroids or any other form of immunosuppressive therapy within 7 days prior to start of study drug.
7. History of autoimmune diseases requiring systemic immunosuppressive therapy in the last 2 years
8. Pregnant or nursing women.
9. Treatment with radiation therapy, major surgery, chemotherapy, or investigational therapy within 4 weeks prior to study entry (6 weeks for nitrosoureas or mitomycin C). Radiation for palliation of pain is allowed within 1 week prior to study entry, but the lesion should not be selected as a target lesion for RECIST analysis.
10. Unwillingness or inability to comply with procedures required in this protocol
11. Known active infection with human immunodeficiency virus (HIV), human T-cell leukemia virus, type 1 (HTLV-1), hepatitis B virus (HBV), or hepatitis C virus (HCV)

    * Patients with a history of hepatitis B or C are allowed if HBV DNA or HCV RNA are undetectable
    * Active infection with HIV and CD4+ T-cell count <350/μL. Patients not on established anti-retroviral therapy for at least 4 weeks and having a detectable HIV viral load
12. Serious uncontrolled nonmalignant disease (e.g., renal failure, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the investigator and/or the sponsor
13. Prior treatment with an IL-2 targeted treatment, unless given as a part of a tumor infiltrating lymphocyte treatment combination;
14. Known sensitivity to IL-2 or any of the excipients in ODC-IL2;
15. Active treatment with heparin or heparin-related therapies, unless the patient can be transitioned to a non-heparin treatment for the clinical condition with an adequate washout prior to enrollment in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) | 28 days
Incidence of Treatment-Emergent Adverse Events (TEAEs) | From the first administration of study drug, throughout the course of the study, and for 90 days after the last dose of study drug
  All AEs will be assessed per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 and American Society for Transplantation and Cellular Therapy (ASTCT) Consensus Grading for cytokine release syndrome (CRS) based on investigator assessment.
Incidence of changes in clinical laboratory abnormalities | From the first administration of study drug, throughout the course of the study, and for 90 days after the last dose of study drug

SECONDARY OUTCOMES:
Serum concentrations of ODC-IL2, free IL-2 and drug backbone following release of IL-2 | 24 months
Investigator-assessed Objective response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | 24 months
Disease control rate (DCR) by RECIST 1.1 | through 6 months after start of treatment
Duration of response (DoR) by RECIST 1.1 | 24 months
Progression-free survival (PFS) by RECIST 1.1 | 24 months
To assess tumor biopsies for pharmacodynamic markers of target engagement and immune pathway activation | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- HonorHealth, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
The individual participant study data and trial results will be shared with the study Investigators and the FDA, as well as presented and/or published in medical journals and conferences.